CLINICAL TRIAL: NCT04163718
Title: A Phase 2 Study to Assess the Efficacy, Safety, Pharmacokinetic and Pharmacodynamic Parameters of Umbralisib in Treatment Naïve Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: TGR-1202 (Umbralisib) in Treatment Naïve Patients With Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug no longer available
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19585; TGR-1202-203 (Other: TG Therapeutics, Inc.)
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with Umbralisib (Experimental)
  Interventions: Drug: Umbralisib

INTERVENTIONS:
Drug: Umbralisib — 800 mg Umbralisib will be self-administered on an outpatient basis. Umbralisib will be taken orally once daily within 30 minutes of a meal until removal from study. This treatment will be administered in 4 week (28-day) cycles.
  Other Names: TGR-1202

SUMMARY:
The purpose of this study is to see how safe and effective the investigational drug umbralisib (TGR-1202) is in individuals with Chronic Lymphocytic Leukemia (CLL)

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of B-cell CLL that has not been previously treated and now warrants treatment consistent with accepted iwCLL criteria (Hallek 2018) for initiation of therapy. Any one of the following conditions constitute CLL that warrants treatment: (a) Evidence of progressive marrow failure as manifested by the onset or worsening of anemia and/or thrombocytopenia, or (b) Massive (i.e., lower edge of spleen ≥ 6 cm below the left costal margin), progressive, or symptomatic splenomegaly, or (c) Massive (i.e., ≥ 10 cm in the longest diameter), progressive, or symptomatic lymphadenopathy, or (d) Progressive lymphocytosis in the absence of infection, with an increase in blood absolute lymphocyte count (ALC) >50% over a 2-month period or lymphocyte doubling time of <6 months (as long as initial ALC was ≥30,000/µL), or e) Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy, or (f) Symptomatic or functional extranodal involvement (e.g. skin, kidney, lung, or spine), or (g) Constitutional symptoms, defined as any one or more of the following disease-related symptoms or signs occurring in the absence of evidence of infection: (i) Unintentional weight loss of ≥10% within the previous 6 months, or (ii) Significant fatigue (≥ Grade 2), or (iii) Fevers >100.5°F or 38.0°C for ≥2 weeks, or (iv) Night sweats for >1 month.
* Adequate organ system function as defined per protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Ability to swallow and retain oral medication
* Female participants who are not of child-bearing potential and female participants of child-bearing potential who have a negative serum pregnancy test within 3 days prior to Cycle 1, Day 1. Female participants of child-bearing potential and all male partners, and male participants must consent to use a medically acceptable method of contraception throughout the study period and for 30 days after the last dose of study drug.
* Willingness and ability to comply with trial and follow-up procedures, and give written informed consent

Exclusion Criteria:

* Has ever received any form of treatment for CLL.
* Corticosteroid therapy of prednisone > 10 mg or equivalent started at least 7 days prior to Cycle 1, Day 1 is prohibited. Prednisone ≤ 10 mg daily or equivalent is allowed as clinically warranted. Topical or inhaled corticosteroids are permitted.
* Prior treatment with umbralisib.
* Prior treatment with autologous hematologic stem cell transplant or prior Allogeneic hematologic stem cell transplant is excluded.
* Evidence of chronic active Hepatitis B (HBV, not including participants with prior hepatitis B vaccination; or positive serum Hepatitis B antibody) or chronic active Hepatitis C infection (HCV), active cytomegalovirus (CMV), or known history of HIV.
* Known histological transformation from CLL to an aggressive lymphoma (i.e. Richter's transformation / Hodgkin Lymphoma).
* Evidence of ongoing systemic bacterial, fungal or viral infection, except localized fungal infection of skin/nails. NOTE: Participants may be receiving prophylactic antiviral or antibacterial therapies at investigator discretion. Use of anti-pneumocystis and antiviral prophylaxis is required.
* Inflammatory bowel disease (such as Crohn's disease or ulcerative colitis)
* Malabsorption syndromes
* Irritable bowel syndrome with greater than 3 loose stools per day as a baseline.
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:(a) Symptomatic, or history of documented congestive heart failure (NY Heart Association functional classification III-IV) - See Appendix B (b) Myocardial infarction within 6 months of enrollment (c) Concomitant use of medication known to cause QT prolongation or torsades de pointes should be used with caution and at investigator discretion. (d) Angina not well-controlled by medication (e) Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), symptomatic peripheral arterial disease, angioplasty, cardiac/vascular stenting within 6 months of enrollment.
* Malignancy, including myelodysplastic syndromes, within 3 years of study enrollment except for basal, squamous cell carcinoma or melanoma in situ, carcinoma in situ of the cervix, superficial bladder cancer not treated with intravesical chemotherapy or Bacillus Calmette-Guerin (BCG) within 6 months, localized prostate cancer following curative treatment and with a normal PSA.
* Women who are pregnant or lactating.
* Participants requiring immediate cytoreductive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pinilla, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Umbralisib
Started | 12
Completed | 0
Not Completed | 12
Not completed — Study terminated | 12

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Umbralisib
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Response and Partial Response)
Description: Overall Response Rate (ORR) of Umbralisib Treatment will be determined according to the criteria of the International Workshop on Chronic Lymphocytic Leukemia. ORR is defined as the percent of participants who achieve Complete Response (CR) or Partial Response (PR). Due to early study termination, result data is provided as best response at End of Treatment/Study Termination.
Time Frame: Up to 24 months
Population: Evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Umbralisib
Number analyzed (Participants) | 9
Participants
  Stable Disease | 1
  Partial Response | 8

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as the interval from registration to the earlier of the first documentation of definitive disease progression or death from any cause.
Time Frame: Up to 24 months
Population: PFS cannot be calculated. Drug was withdrawn by FDA, therefore all participants off treatment too early to determine survival.
Measure: Number; unit: participants
Arm/Group | Treatment With Umbralisib
Number analyzed (Participants) | 9
participants | NA — Insufficient number of participants with events because drug was withdrawn by FDA, therefore all participants off treatment too early

3. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants with adverse events after receiving one dose of Umbralisib..
Time Frame: Up to 15 months
Measure: Number; unit: participants
Arm/Group | Treatment With Umbralisib
Number analyzed (Participants) | 12
participants | 10

ADVERSE EVENTS:
Time Frame: Adverse events collected from on treatment date through off study date, an average of 15 months.
Arm/Group | Treatment With Umbralisib
All-Cause Mortality (participants affected / at risk) | 2/12
Serious Adverse Events (participants affected / at risk) | 10/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Umbralisib (N=12)
Fever (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Death, NOS (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COVID-19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — lung adenocarcinoma
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 1 (1)
Musculoskeletal and connective tissue disorder-Other (Musculoskeletal and connective tissue disorders) | 1 (1) — broken hip
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cardiac disorders -Other (Cardiac disorders) | 1 (1) — left bundle branch block
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2)
General disorders and administration site conditions -Other (General disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Umbralisib (N=12)
Nausea (Gastrointestinal disorders) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 7 (13)
Bloating (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (15)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 3 (5)
Alanine aminotransferase increased (Investigations) | 2 (3)
Weight loss (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (2)
Dysgeusia (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3)
Concentration impairment (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Akathisia (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Pain (General disorders) | 5 (8)
Fever (General disorders) | 3 (4)
Edema limbs (General disorders) | 2 (4)
Fatigue (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (9)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 3 (3)
Eye infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Confusion (Psychiatric disorders) | 3 (5)
Anxiety (Psychiatric disorders) | 2 (3)
Hallucinations (Psychiatric disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (4)
Flushing (Vascular disorders) | 2 (4)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT04163718/Prot_SAP_000.pdf